CLINICAL TRIAL: NCT02459782
Title: Ultrasound Guided Peribulbar Anaesthesia: a Real-time Ultrasound Guided Technique With a Novel Dual Quadrant Injection
Brief Title: Ultrasound Guided Peribulbar Anaesthesia - A Novel Dual Quadrant Injection Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 424-2011
Record Dates: First submitted 2015-03-20; First posted 2015-06-02 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-05

CONDITIONS: Eye Diseases
Keywords: Ultrasound guided peribulbar anesthesia
MeSH Terms: conditions — Eye Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- US Guided Dual Quadrant Peribulbar block (Other): Ultrasound guided Dual Quadrant Peribulbar Anaesthesia
  Interventions: Procedure: Ultrasound guided Dual Quadrant Peribulbar Anaesthesia

INTERVENTIONS:
Procedure: Ultrasound guided Dual Quadrant Peribulbar Anaesthesia — Landmark Guided single injection vs Ultrasound guided dual quadrant injection

SUMMARY:
Peribulbar anaesthesia for ocular surgery depends on the spread of local anaesthetic throught the orbit to be successful and has a relatively high failure rate. This study will examine a novel ultrasound guided approach to peribulbar anaesthesia which should extend the depostion of local anaesthetic by using a dual quadrant injection technique. The study will assess the feasibility of this technique, how successful it is and whether any obvious safety issues arise with its use.

DETAILED DESCRIPTION:
Peribulbar anesthesia is widely used for anterior and posterior chamber ophthalmic procedures. It is a blind technique which is traditionally carried out by inserting a needle in the infero-lateral aspect of the orbit below the globe and injecting a volume of 8 - 12 mL of local anesthetic in the periorbital space. The goal of this inejction is to achieve akinesia and anesthesia of the eye sufficient for surgery. The technique has a relatively high failure rate of up to 30%. A failure or insufficient block requires a second or rarely a third peribulbar injection to achieve success. Ultrasound can be used to guide needles in the human body and has been successfully used in many anatomic locations for anaesthesia. This study will assess whether ultrasound can guide the block needle in ophthalmic anesthesia to deliver local anesthetic via a single entry into two discrete locations within the periorbital space - the first in the infero-lateral quadrant and the second in the infero-medial quadrant. If this can be done the investigators may achieve a higher success rate for this block with a lower volume potentially improving the quality of the block and its safety.

ELIGIBILITY:
Inclusion Criteria:

* ASA score less than III and ability to provide a written informed consent
* 22 patients presenting for opthalmic surgery

Exclusion Criteria:

* Coagulation disorder or anticoagulated with INR > 1.5
* Platelet count < 75 X 10*9/L
* Significant Myopia (axial length > 28mm)
* Patients unable to lie supine for 2 hours
* Patients with recent gas or silicone injections in/around the eye

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-01; Primary Completion 2012-03 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Block Success | 10 minutes post intervention
  Block will be deemed a failure if a supplementary block is required for the operative procedure

SECONDARY OUTCOMES:
Block Quality (standardized Ocular Scoring System for akinesia and anaesthesia) | 5 and 10 minutes
  Block will be assessed according to a standardized Ocular Scoring System for akinesia and anaesthesia at 5 minutes and 10 minutes post block. This is a composite measure
Block Volume | 1 minute
  Total volume of local anaesthetic will be recorded. Volume for each part of the dual injection technique will also be recorded. This is a composite measure.
Duration of Procedure | 1 to 10 minutes
  The duration of the entire procedure will be recorded
Complications | 6 Weeks
  Any complications during the procedure or in follow up clinical visits will be recorded
Image Visualization | 1 minute
  Operator's ability to see the needle in both the infero-lateral and infero-medial injection will be recorded. Ability to see perineural, retrobulbar and medial rectus spread of local anaesthetic will be recorded. This is a composite qualitative measure.

CONTACTS AND LOCATIONS:
Overall Officials: Paul G McHardy, MD, Principal Investigator — Sunnybrook Health Sciences Centre